CLINICAL TRIAL: NCT06357806
Title: The Safety and Efficacy of PD-1 Antibody Combined With Pegylated Interferon-α Therapy to Promote the Clinical Cure in Nucleoside (Acid) Analogues-suppressed Chronic Hepatitis B Patients: A Protocol for the Prospective Pilot Study
Brief Title: The Treatment of PD-1 Antibody Combined With Peg-IFNα in NAs-suppressed CHB Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIN-CHB-1
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — sintilimab; nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peg-IFNα group (Active Comparator): 180 ug Peg-IFNα-2b subcutaneous injection once/week for 48 weeks NAs
  Interventions: Drug: Peg-IFNα-2b; Drug: NAs
- PD-1 antibody group (Active Comparator): 1.5 mg/kg Sintilimab intravenous injection once per 3 weeks for 24 weeks NAs
  Interventions: Drug: Sintilimab; Drug: NAs
- PD-1 antibody combined Peg-IFNα group (Experimental): 1.5 mg/kg Sintilimab intravenous injection once per 3 weeks for 24 weeks 180 ug Peg-IFNα-2b subcutaneous injection once/week for 48 weeks NAs
  Interventions: Drug: Sintilimab; Drug: Peg-IFNα-2b; Drug: NAs

INTERVENTIONS:
Drug: Sintilimab — 100mg/10ml/1bottle
  Arms: PD-1 antibody combined Peg-IFNα group; PD-1 antibody group
Drug: Peg-IFNα-2b — 180ug/0.5ml/1bottle
  Arms: PD-1 antibody combined Peg-IFNα group; Peg-IFNα group
Drug: NAs — tablets
  Other Names: ETV/TDF/TAF

SUMMARY:
This is a prospective, open-labled, randomized controlled study to assess efficacy and safety of treatment with Sintilimab (PD-1 antibody) combined Peg-IFNα-2b in CHB patients on stable NAs treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years old;
2. Chronic hepatitis B patients with clear diagnosis of hematology, etiology and clinical (for example: HBsAg positive for more than 6 months);
3. Treatment with NAs (ETV, TDF or TAF）at least 1 years and continue NAs therapy during screening;
4. HBV DNA and HBeAg turn negative after NAs treatment;
5. HBsAg ranged 200-1000 IU/ml.

Exclusion Criteria:

1. Cirrhosis;
2. platelet count < 90×10^9/L, WBC count < 3.0×10^9/L, neutrophil count < 1.3×10^9/L, ALT > ULN（40U/L）, total bilirubin > 2ULN;
3. History of or suspicion of hepatocellular carcinoma
4. Patients received interferon therapy within 12 months;
5. Patients received immunosuppressive therapy or other therapy influenced study within 12 months;
6. Hepatitis A, hepatitis C, hepatitis D, HIV infection or other active infections;
7. Alcohol or drug abuse/dependence;
8. Investigator judges that the participants are not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
The rate of HBsAg loss at 24 weeks and 48 weeks. | 48 weeks
  Evaluate the level of HBsAg at 24 weeks and 48 weeks.
Incidence of treatment-emergent adverse events/serious adverse events | 48 weeks
  Evaluate the treatment-emergent adverse events/serious adverse events

SECONDARY OUTCOMES:
The rate of HBsAg decline > 1log(IU/ml) at 24 weeks and 48 weeks | 48 weeks
  Evaluate the level of serum HBsAg at 24 weeks and 48 weeks.
The rate of HBsAb positive at 24 weeks and 48 weeks. | 48 weeks
  Evaluate the level of serum HBsAb at 24 weeks and 48 weeks.
The concentration of HBcrAg at baseline, 12 weeks, 24 weeks and 48 weeks. | 48 weeks
  Evaluate the level of serum HBcrAg at baseline, 12 weeks, 24 weeks and 48 weeks.
The concentration of pgRNA at baseline, 12 weeks, 24 weeks and 48 weeks. | 48 weeks
  Evaluate the level of serum pgRNA at baseline, 12 weeks, 24 weeks and 48 weeks.
The concentration of anti-HBc at baseline, 12 weeks, 24 weeks and 48 weeks. | 48 weeks
  Evaluate the level of serum anti-HBc at baseline, 12 weeks, 24 weeks and 48 weeks.
Immune response of T cell, B cell, NK cell at baseline, 12 weeks, 24 weeks and 48 weeks. | 48 weeks
  Evaluate the frequency and function of T cell, B cell, NK cell (tested by flowcytometry/fluorospot/elispot)

CONTACTS AND LOCATIONS:
Locations (1):
- the Fifth Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Li X, Lu J, Zhang X, Dang S, Li Y, He Y, Guo Y, Wang J, Maimaitijiang W, Zheng S, Ren S, Cao H, Zhang W, Zhang X, Ma H, Wang FS, Fu J. Safety and efficacy of PD-1 antibody combined with pegylated interferon alpha for functional cure in nucleos(t)ide analogues-suppressed chronic hepatitis B patients: protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Sep 21;15(9):e105710. doi: 10.1136/bmjopen-2025-105710. PMID 40976664